CLINICAL TRIAL: NCT01462006
Title: Double-blind Placebo-controlled Pilot Study of Sirolimus in IPF
Brief Title: Double-blind Placebo-controlled Pilot Study of Sirolimus in Idiopathic Pulmonary Fibrosis (IPF)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Borna Mehrad, MD, Professor, Department of Medicine, Pulmonary and Critical Care, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15282; R01HL098329 (NIH)
Record Dates: First submitted 2011-10-26; First posted 2011-10-28 (Estimated); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Idiopathic Pulmonary Fibrosis; Diffuse Parenchymal Lung Disease; Interstitial Lung Disease
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Lung Diseases, Interstitial | interventions — Sirolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sirolimus (Experimental)
  Interventions: Drug: sirolimus
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: sirolimus — randomized to drug or placebo, followed by washout, followed by crossover
  Arms: Sirolimus
Other: Placebo — randomized to drug or placebo, followed by washout, followed by crossover
  Arms: Placebo

SUMMARY:
Idiopathic pulmonary fibrosis (IPF) is an illness characterized by progressive decline in lung function and premature death from respiratory failure. Fibrocytes are a novel population of bone marrow-derived circulating progenitor cells that have been shown to traffic to the lungs and contribute to fibrosis in animal models of pulmonary fibrosis, and whose numbers correlate with the degree of fibrosis and with survival in human pulmonary fibrosis. The investigators propose to test the hypothesis that therapy with the mTOR inhibitor, sirolimus, reduces the number of circulating fibrocytes in patients with IPF. The investigators propose to test this hypothesis in short-term pilot trial of sirolimus in patients with IPF to determine its effect on the number and phenotype of circulating fibrocytes.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients 21-85 years of age
2. Individuals diagnosed with IPF, based on:

   * clinical symptoms consistent with idiopathic pulmonary fibrosis (IPF) of > 3 months duration, plus
   * histologically diagnosed UIP or diagnostic chest high resolution CT features of UIP, plus
   * negative workup for known causes of UIP
3. Ability to understand a written informed consent form and comply with the requirements of the study.

Exclusion Criteria:

1. Clinical features or known diagnosis of an active infection, including untreated latent tuberculosis
2. Clinical features or known diagnosis of malignancy
3. Known diagnosis of an interstitial lung disease other than IPF including but not limited to sarcoidosis, hypersensitivity pneumonitis, non-specific interstitial pneumonia (NSIP).
4. History of clinically significant environmental exposures known to cause interstitial lung disease (including but not limited to drugs, asbestos, silica, beryllium, radiation, domestic birds, etc).
5. Diagnosis of any connective tissue disease (including but not limited to scleroderma, SLE, rheumatoid arthritis) or vasculitides according to the American College of Rheumatology criteria.
6. Systolic blood pressure < 100 or >145 mm Hg or diastolic blood pressure < 50 or >90 mmHg
7. Evidence of active infection within 1 week prior to enrollment.
8. Recently started (<8 weeks prior to baseline visit) or planned cardiopulmonary rehabilitation program before conclusion of the study
9. History of unstable or deteriorating cardiac disease, including but not limited to: myocardial infarction, coronary artery bypass surgery or angioplasty within the past 6 months, congestive heart failure requiring hospitalization within the past 6 months, or uncontrolled arrhythmia
10. History of unstable or deteriorating neurologic disease, including but not limited to: TIAs or stroke
11. Pregnant or lactating females. Females of child bearing potential are required to have a negative serum or urine pregnancy test prior to treatment and agree to practice abstinence or prevent pregnancy by at least a barrier method of birth control.
12. Liver panel above specific limits at screening: Total bilirubin >1.5-fold upper limit of normal, AST, ALT or alkaline phosphatase > 3-fold upper limit of normal at screening.
13. Hematology outside of specified limits, WBC <2,500/ mm3, hematocrit <30, platelets <100,000/mm3 at screening.
14. Investigational therapy for any indication within 28 days prior to treatment.
15. Current treatment with drugs that are strong inhibitors of CYP3A4 or P-gp, namely bromocriptine, cimetidine, cisapride, clotrimazole, danazol, diltiazem, fluconazole, HIV-protease inhibitors (e.g., ritonavir, indinavir), metoclopramide, nicardipine, troleandomycin, verapamil
16. Inability or unwillingness to comply with the requirements for the trial.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
fibrocytes | up to 22 weeks
  change in peripheral blood concentration of CXCR4+ fibrocytes
number of subjects with drug side-effects | up to 22 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Borna Mehrad, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Derived] Gomez-Manjarres DC, Axell-House DB, Patel DC, Odackal J, Yu V, Burdick MD, Mehrad B. Sirolimus suppresses circulating fibrocytes in idiopathic pulmonary fibrosis in a randomized controlled crossover trial. JCI Insight. 2023 Apr 24;8(8):e166901. doi: 10.1172/jci.insight.166901. PMID 36853800